CLINICAL TRIAL: NCT05930093
Title: Multi-center, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of LivPhcD Capsules in the NAFLD Subjects
Brief Title: Evaluate the Efficacy and Safety of LivPhcD Capsules in the NAFLD Subjects
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: TCM Biotech International Corp. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LivPhcD-001
Record Dates: First submitted 2023-05-28; First posted 2023-07-05 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: NAFLD
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Placebo (Placebo Comparator): Placebo without active ingredient
  Interventions: Dietary Supplement: Placebo
- 2 cap.LivPhcD/per day (Active Comparator): 515mg/LivPhcD cap. 2 cap./per day
  Interventions: Dietary Supplement: 2 cap.LivPhcD/per day
- 4 cap.LivPhcD/per day (Active Comparator): 515mg/LivPhcD cap. 4 cap./per day, BID
  Interventions: Dietary Supplement: 4 cap.LivPhcD/per day
- 6 cap.LivPhcD/per day (Active Comparator): 515mg/LivPhcD cap. 6 cap./per day, TID
  Interventions: Dietary Supplement: 6 cap.LivPhcD/per day

INTERVENTIONS:
Dietary Supplement: Placebo — Placebo matching LivPhcD cap.
  Arms: Placebo
Dietary Supplement: 2 cap.LivPhcD/per day — 2 caps. LivPhcD cap. after meal, once a day
  Arms: 2 cap.LivPhcD/per day
Dietary Supplement: 4 cap.LivPhcD/per day — 4 caps. LivPhcD cap. after meal, BID
  Arms: 4 cap.LivPhcD/per day
Dietary Supplement: 6 cap.LivPhcD/per day — 6 caps. LivPhcD cap. after meal, TID
  Arms: 6 cap.LivPhcD/per day

SUMMARY:
Non-alcoholic fatty liver disease (also called NAFLD) is a disease in which excessive fat accumulates in the liver of a patient without a history of alcohol abuse. Early-stage NAFLD does not usually cause any harm but nonalcoholic steatohepatitis (NASH) can lead to serious liver damage, including fibrosis or cirrhosis. Nearly 25% of the world's population is affected by NAFLD.

There are no FDA-approved medications for the treatment of NAFLD currently and although lifestyle modifications with appropriate diet and exercise have been shown to be beneficial, this has been difficult to achieve and sustain for the majority of patients.

LivPhcD™ capsule have shown hepatoprotective effects in both animal and human data. This study aims to investigate the effects of LivPhcD™ capsule in hepatocellular lipid content using Fibroscan.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female between 20 and 75 years of age.
2. Capable of giving written informed consent and able to effectively communicate with the investigator and study personnel.
3. Has a body mass index (BMI) ≥20 kg/m^2 and ≤50 kg/m^2 and stable weight for the past 3 months
4. CAP ≥ 238 db/m
5. Fibro scan (transient elastography) F0~F3

Exclusion Criteria:

1. Pregnant or breastfeeding or planning to become pregnant or unwilling to use an acceptable contraceptive method to avoid pregnancy during the study period
2. Type 1 diabetes mellitus.
3. History of other causes of chronic liver disease [autoimmune, primary biliary cirrhosis, HBV (HBsAg positive) and HCV, Wilson disease, alpha-1-antitrypsin deficiency, hemochromatosis etc.
4. Use of medications that could induce steatosis, such as estrogen or other hormonal replacement therapy, amiodarone, methotrexate, tamoxifen, raloxifene, pharmacological doses of oral glucocorticoids (≥10 mg per day of prednisone or equivalent), or chloroquine.
5. Use of vitamin E (doses ≥800 IU/dy) or pioglitazone or SGLT2 inhibitor or GLP-1 agonists any FDA-approved drug for NASH to be approved during the study.
6. Has significant systemic or major illnesses other than liver disease, ex: recent events (≤6 months before study entry) of congestive heart failure, unstable coronary artery disease, serious COPD, renal failure and need hemodialysis, stroke, transient ischemic attack, or organ transplantation
7. Known alcohol abuse or alcohol use disorder (>20 g/day for women; >30 g/day for men)
8. Has the abnormal data including: fasting TG >400 mg/dL ; ALT or GGT>5.0 x ULN；Bilirubin >2 x ULN，unless due to an alternative etiology such as Gilbert's syndrome; INR ≥1.3; Albumin < LLN; Platelet <0.95x LLN
9. Subjects with hemoglobin A1c (HbA1c) >8.5% within 3 months before study entry
10. Plan to have major surgery during the study period (bariatric surgery, biliary diversion surgery)
11. Participation in any other investigational clinical trial within 30 days of entry to this protocol(including drugs, medical devices, novel medical technologies, food, and lifestyle interventions affecting diet, exercise, and circadian rhythm investigational clinical trial.);
12. History of HIV

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2023-12-07 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Reduction of Liver Fat | 36 weeks
  Between group difference in the proportion of patients with ≥ 10% reduction of baseline of liver fat by CAP(Controlled Attenuation Parameter)

SECONDARY OUTCOMES:
Change in liver fat at least 30% reduction | 24 weeks and 36 weeks
  Between group difference in the proportion of patients with ≥ 30% reduction of baseline of liver fat by CAP
Change in liver fat at least 1 stage reduction | 24 weeks and 36 weeks
  Between group difference in the proportion of patients with 1 stage reduction of baseline of liver fat by CAP
Change in liver fat | 24 weeks and 36 weeks
  Between group difference in mean change of liver fat by CAP
Stable in liver fat | 24 weeks and 36 weeks
  Between group difference in the proportion of patients with stable of baseline of liver fat by CAP
Change in liver fibrosis at least 10% reduction | 24 weeks and 36 weeks
  Between group difference in the proportion of patients with ≥ 10% reduction of baseline of liver fibrosis by Fibroscan
Change in liver fibrosis at least 1 stage reduction | 24 weeks and 36 weeks
  Between group difference in the proportion of patients with 1 stage reduction of baseline of liver fibrosis by Fibroscan
Stable in liver fibrosis | 24 weeks and 36 weeks
  Between group difference in the proportion of patients with stable reduction of baseline of liver fibrosis by Fibroscan
Change in liver fibrosis | 24 weeks and 36 weeks
  Between group difference in mean change of FIB-4
Change in ALT | 24 weeks and 36 weeks
  Between group difference in mean change or in the proportion of patients of ALT
Change in AST | 24 weeks and 36 weeks
  Between group difference in mean change or in the proportion of patients of AST
Change in GGT | 24 weeks and 36 weeks
  Between group difference in mean change or in the proportion of patients of GGT
Change in AP | 24 weeks and 36 weeks
  Between group difference in mean change or in the proportion of patients of AP
Change in Bilirubin | 24 weeks and 36 weeks
  Between group difference in mean change or in the proportion of patients of Bilirubin
Change in Triglyceride | 24 weeks and 36 weeks
  Between group difference in mean change or in the proportion of patients of Triglyceride
Change in Total Cholesterol | 24 weeks and 36 weeks
  Between group difference in mean change or in the proportion of patients of Total Cholesterol
Change in HDL-C | 24 weeks and 36 weeks
  Between group difference in mean change or in the proportion of patients of HDL-C
Change in LDL-C | 24 weeks and 36 weeks
  Between group difference in mean change or in the proportion of patients of LDL-C
Change in TNF-α | 24 weeks and 36 weeks
  Between group difference in mean change or in the proportion of patients of TNF-α
Change in C-Reactive Protein | 24 weeks and 36 weeks
  Between group difference in mean change or in the proportion of patients of C-Reactive Protein
Change in Albumin | 24 weeks and 36 weeks
  Between group difference in mean change or in the proportion of patients of Albumin
Occurrence of adverse events and serious adverse events | 24 weeks and 36 weeks
  Between group difference in the occurrence of adverse events and serious adverse events.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Not Required For This Country, Taiwan